CLINICAL TRIAL: NCT07222852
Title: Cardiovascular Protection After Preeclampsia With Enalapril
Acronym: CAPP-E
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2310266-3
Record Dates: First submitted 2025-10-02; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Preeclampsia; Hypertensive Disorder of Pregnancy; Hypertension; Gestational Hypertension; Gestational Hypertension After Childbirth
Keywords: postpartum hypertension, preeclampsia, gestational hypertension
MeSH Terms: conditions — Pre-Eclampsia; Toxemia; Hypertension; Hypertension, Pregnancy-Induced | interventions — Enalapril

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Enalapril (Experimental): First-line anti-hypertensive treatment with enalapril
  Interventions: Drug: Enalapril
- Standard treatment (Active Comparator): First-line anti-hypertensive treatment with standard of care treatment
  Interventions: Other: Standard treatment

INTERVENTIONS:
Drug: Enalapril — First-line anti-hypertensive treatment with enalapril
  Arms: Enalapril
Other: Standard treatment — First-line anti-hypertensive treatment per standard of care
  Arms: Standard treatment

SUMMARY:
The purpose of this study is to learn if postpartum women are willing to be randomized to different blood pressure medicines after delivery and how that affects blood pressure in women with hypertensive disorders of pregnancy.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in women worldwide, and despite declines in all other age groups, mortality rates attributed to CVD are increasing in women of childbearing age. Hypertensive disorders of pregnancy (HDP), including preeclampsia and gestational hypertension, are well-established risk factors for CVD across diverse patient populations. There is compelling evidence that the preponderance of HDP-associated CVD risk is linked to progression to chronic hypertension following pregnancy. Thus, the postpartum period after HDP is a critical yet under-studied opportunity for intervention to prevent chronic disease in women.

One intervention that may reduce the chance of progression to CVD is the institution of anti-hypertensive medications. The cornerstones of current postpartum anti-hypertensive treatment are labetalol (a dual β- and α-adrenergic receptor blocker) and nifedipine (a calcium channel blocker), primarily due to their well-documented safety profile during pregnancy and obstetricians' comfort with their dosing. However, there are significant limitations in the current standard of care for anti-hypertensive treatment postpartum, including (1) two to three times per day dosing, (2) significant side effects, and (3) lack of endothelial or cardioprotective effects. Further, there is some evidence that these medications may not be as efficacious as some others.

Angiotensin-converting enzyme (ACE) inhibitors are anti-hypertensive agents that provide cardioprotection through anti-inflammatory effects, increased nitric oxide bioavailability, and diminished fibrosis. Because of these benefits, they are recommended in non-pregnant / postpartum individuals who have heart failure or myocardial infarction to reduce cardiovascular mortality. Enalapril is a type of ACE- inhibitor that is taken daily or twice daily with minimal side effects, is a highly effective anti-hypertensive agent, and has a reassuring lactation safety profile, making it an ideal candidate for postpartum treatment after preeclampsia.

The overall objective of this application is to conduct a single-site RCT, which will enroll individuals within the institution's remote blood pressure (BP) management program, to allow the collection of key data that will inform a future NIH-funded RCT. The' central hypothesis is that an RCT evaluating enalapril versus standard-of-care treatments will be feasible, and that enalapril will improve blood pressure at 4 months after delivery. The investigators will test this hypothesis by pursuing the following specific aims:

Aim 1. Determine the feasibility of conducting a randomized controlled trial of enalapril versus current standard of care (labetalol or nifedipine) in postpartum individuals who have had a hypertensive disorder of pregnancy.

Aim 2. Determine whether enalapril versus standard of care improves blood pressure at 4 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum individuals
* ≥18 years old
* Hypertensive disorder of pregnancy
* Enrolled in Women and Infants Hospital Hypertension Equity remote monitoring program.

Exclusion Criteria:

* Maternal cardiac disease
* Individuals with pre-pregnancy hypertension or diabetes
* Allergy or contraindication to enalapril

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enrollment | 4 months
  Proportion of approached individuals who are enrolled
Feasibility of retention | 4 months
  Retention of participants to 4 months postpartum

SECONDARY OUTCOMES:
Blood pressure | 4 months
  Systolic and diastolic blood pressure
Blood pressure | 6 weeks
  Systolic and diastolic blood pressure
Mean home blood pressure | 6 weeks
  Mean systolic and diastolic blood pressure
Mean arterial pressure | 4 months
  Mean arterial blood pressure
Mean arterial pressure | 6 weeks
  Mean arterial blood pressure
Quantification of anti-hypertensive agents through study period using therapeutic intensity score | 4 months
  Throughout study period
Use of anti-hypertensive agents | 4 months
  At study completion
Medication side effects | 4 months
  Throughout study period

CONTACTS AND LOCATIONS:
Overall Officials: Alisse Hauspurg, MD, Principal Investigator — WOMEN AND INFANTS HOSPITAL-RHODE ISLAND

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after publication of primary manuscript